CLINICAL TRIAL: NCT03182907
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of a Single Infusion of Bezlotoxumab (MK-6072, Human Monoclonal Antibody to C. Difficile Toxin B) in Children Aged 1 to <18 Years Receiving Antibacterial Drug Treatment for C. Difficile Infection (MODIFY III)
Brief Title: Bezlotoxumab (MK-6072) Versus Placebo in Children With Clostridium Difficile Infection (CDI) (MK-6072-001)
Acronym: MODIFY III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 6072-001; MK-6072-001 (Other: Merck); 2017-000070-11 (EudraCT Number)
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Results first posted 2023-06-07 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — bezlotoxumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bezlotoxumab (Experimental): Participants receive 10 mg of bezlotoxumab per kg body weight via a single 60-minute (±10 minutes) intravenous (IV) infusion on Day 1. Additionally, participants receive background antibacterial drug treatment (ABD) for 10-21 days per institutional guidelines, at the investigator's discretion. Dose may then be changed based on results from initial 12 participants.
  Interventions: Biological: Bezlotoxumab; Drug: Antibacterial drug treatment (ABD)
- Placebo (Placebo Comparator): Participants receive placebo for bezlotoxumab consisting of either 0.9% sodium chloride or 5% dextrose via a single 60-minute (±10 minutes) IV infusion on Day 1. Additionally, participants receive background ABD for 10-21 days per institutional guidelines, at the investigator's discretion.
  Interventions: Drug: Placebo; Drug: Antibacterial drug treatment (ABD)

INTERVENTIONS:
Biological: Bezlotoxumab — A single intravenous (IV) infusion of 10 mg of bezlotoxumab per kg body weight. Dose may then be changed based on results from initial 12 participants.
  Other Names: MK-6072
  Arms: Bezlotoxumab
Drug: Placebo — A single IV infusion of placebo for bezlotoxumab consisting of either 0.9% sodium chloride or 5% dextrose.
  Arms: Placebo
Drug: Antibacterial drug treatment (ABD) — ABD will be administered for 10-21 days including the duration of ABD prior to the screening visit, during the screening period, and after the infusion of study treatment, per institutional guidelines, at the investigator's discretion. ABD is defined as the receipt of oral metronidazole, oral vancomycin, intravenous (IV) metronidazole concurrent with oral vancomycin, oral fidaxomicin, or oral fidaxomicin concurrent with IV metronidazole.

SUMMARY:
The primary objectives of this study are to evaluate the pharmacokinetics (PK), safety, and tolerability of bezlotoxumab (MK-6072) in children aged 1 to <18 years of age with a confirmed diagnosis of Clostridium difficile infection (CDI) who are receiving antibacterial drug treatment. The primary hypothesis is that the area under the concentration-time curve from 0 to infinity (AUC0-inf) of bezlotoxumab after treatment of pediatric participants with bezlotoxumab is similar when compared to the AUC0-inf of bezlotoxumab after treatment of adults with bezlotoxumab.

DETAILED DESCRIPTION:
Historical adult pharmacokinetic data is from NCT01241552 and NCT01513239.

ELIGIBILITY:
Inclusion Criteria:

* At screening has suspected or confirmed Clostridium difficile infection (CDI), and is receiving or is planning to receive a 10- to 21-day course of antibacterial drug treatment for CDI
* At study infusion has a diagnosis of CDI confirmed by a diagnostic assay which detects the presence of C. difficile toxin in stool, and is still receiving antibacterial drug treatment for CDI
* Female is not pregnant, and not breastfeeding; but if of childbearing potential agrees to follow contraceptive guidance during the treatment period and for at least 12 weeks after the last dose of study treatment
* Participant and/or parent or caregiver must be able to read, understand, and complete the daily diary

Exclusion Criteria:

* Has an uncontrolled chronic diarrheal illness
* Has a known hypersensitivity to bezlotoxumab, its active substance and/or any of its excipients
* At randomization, their planned course of antibacterial drug treatment for CDI is longer than 21 days
* At screening has received any listed prohibited prior and concomitant treatments and procedures
* Has previously participated in this study, has previously received bezlotoxumab, has received an experimental monoclonal antibody against C. difficile toxin B, or has received a vaccine directed against C. difficile or its toxins.
* Has received an investigational study agent within the previous 30 days, or is currently participating in or scheduled to participate in any other clinical study with an investigational agent during the 12-week study period

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (75):
- United States (21):
  - Children's Hospital - Los Angeles ( Site 0021), Los Angeles, California
  - UCSF Medical Center ( Site 0049), San Francisco, California
  - Children's Hospital - Colorado ( Site 0013), Aurora, Colorado
  - Children's Center for Digestive Healthcare ( Site 0052), Atlanta, Georgia
  - University of Chicago ( Site 0019), Chicago, Illinois
  - Our Lady of the Lake Hospital ( Site 0007), Baton Rouge, Louisiana
  - The Johns Hopkins Rubenstein Child Health Building ( Site 0034), Baltimore, Maryland
  - Tufts Medical Center-Floating Hospital for Children ( Site 0046), Boston, Massachusetts
  - Mayo Clinic - Rochester ( Site 0004), Rochester, Minnesota
  - Washington University ( Site 0037), St Louis, Missouri
  - Columbia University Medical Center/ MSCHONY ( Site 0042), New York, New York
  - SUNY Upstate Medical Center, University Hospital ( Site 0027), Syracuse, New York
  - Montefiore Einstein Center ( Site 0041), The Bronx, New York
  - Duke University Health System ( Site 0025), Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center ( Site 0024), Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center ( Site 0029), Cleveland, Ohio
  - St. Jude Children's Research Hospital ( Site 0050), Memphis, Tennessee
  - Vanderbilt University Medical Center ( Site 0022), Nashville, Tennessee
  - The Children's Hospital of San Antonio ( Site 0009), San Antonio, Texas
  - Primary Children's Hospital ( Site 0001), Salt Lake City, Utah
  - Seattle Childrens Hospital ( Site 0028), Seattle, Washington
- Argentina (2):
  - Hospital Italiano de Buenos Aires. ( Site 2103), Caba, Buenos Aires
  - Hospital Privado de Cordoba ( Site 2102), Córdoba
- Brazil (5):
  - Santa Casa de Misericordia de Belo Horizonte ( Site 0208), Belo Horizonte, Minas Gerais
  - Hospital de Clinicas da Universidade Federal do Parana ( Site 0203), Curitiba, Paraná
  - Hospital Pequeno Principe ( Site 0200), Curitiba, Paraná
  - Hospital Universitario da Universidade Federal de Santa Maria ( Site 0209), Santa Maria, Rio Grande do Sul
  - Instituto de Oncologia Pediatrica - GRAACC - Unifesp ( Site 0205), São Paulo
- Colombia (5):
  - Hospital Pablo Tobon Uribe-Infectology pediatric ( Site 2166), Medellín, Antioquia
  - Fundacion Santa Fe de Bogota ( Site 2167), Bogotá, Bogota D.C.
  - Fundacion Cardioinfantil Instituto de Cardiologia ( Site 2163), Bogotá, Bogota D.C.
  - Fundacion Valle del Lili ( Site 2161), Cali, Valle del Cauca Department
  - Centro Medico Imbanaco ( Site 2160), Cali, Valle del Cauca Department
- Czechia (3):
  - Fakultni Nemocnice Brno Bohunice ( Site 2000), Brno, Brno-mesto
  - Fakultni nemocnice Plzen ( Site 2001), Plzen Lochotin, Plzeň Region
  - 2. LF UK a FN Motol ( Site 2003), Prague
- Germany (2):
  - Universitaetsklinikum Muenster ( Site 1400), Münster, North Rhine-Westphalia
  - Universitaetsklinikum Hamburg Eppendorf ( Site 1402), Hamburg
- Hungary (3):
  - SZTE Szent-Gyorgyi Albert Klinikai Kozpont ( Site 2200), Szeged, Csongrád megye
  - Semmelweis University-II.sz. Gyermekgyógyászati Klinika ( Site 2201), Budapest
  - Del-pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet ( Site 2202), Budapest
- Malaysia (2):
  - Sabah Womens & Childrens Hospital ( Site 3101), Kota Kinabalu, Sabah
  - Hospital Kuala Lumpur ( Site 3100), Kuala Lumpur
- Mexico (4):
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" ( Site 0508), Monterrey, Nuevo León
  - Instituto Tecnologico y de Estudios Superiores de Monterrey ( Site 0502), Monterrey, Nuevo León
  - Instituto Nacional de Pediatria ( Site 0503), Mexico City
  - Hospital Infantil de Mexico Federico Gomez ( Site 0501), Mexico City
- Norway (2):
  - Haukeland universitetssykehus ( Site 1501), Bergen, Vestfold
  - Oslo universitetssykehus ( Site 1500), Oslo
- Poland (5):
  - Wojewodzki Szpital Obserwacyjno Zakazny ( Site 2404), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Instytut Pomnik Centrum Zdrowia Dziecka ( Site 2406), Warsaw, Masovian Voivodeship
  - SPZOZ im. Dzieci Warszawy w Dziekanowie Lesnym ( Site 2405), Łomianki, Masovian Voivodeship
  - Wojewodzki Specjalistyczny Szpital Dzieciecy ( Site 2410), Olsztyn, Warmian-Masurian Voivodeship
  - Wojewodzki Specjalistyczny Szpital im. dr W. Bieganskiego w Lodzi ( Site 2400), Lodz, Łódź Voivodeship
- Portugal (4):
  - Hospital de Braga ( Site 1600), Braga
  - Inst. Portugues de Oncologia de Lisboa Francisco Gentil EPE ( Site 1605), Lisbon
  - Centro Hospitalar de Lisboa Central EPE. Hospital D. Estefania ( Site 1601), Lisbon
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil E.P.E. ( Site 1603), Porto
- Romania (4):
  - Spitalul Clinic de Boli Infectioase Cluj-Napoca ( Site 2502), Cluj-Napoca, Cluj
  - Institutul National de Boli Infectioase Prof. Dr. Matei Bals ( Site 2501), Bucharest
  - Spitalul Clinic de Boli Infectioase si Tropicale Dr. Victor Babes ( Site 2500), Bucharest
  - Spitalul Clinic de Boli Infectioase Constanta ( Site 2504), Constanța
- South Africa (5):
  - Phoenix Pharma Pty Ltd ( Site 2607), Port Elizabeth, Eastern Cape
  - Johese Clinical Research ( Site 2605), Centurion, Gauteng
  - Chris Hani Baragwanath Academic Hospital ( Site 2602), Johannesburg, Gauteng
  - Molotlegi Street ( Site 2603), Pretoria, Gauteng
  - Red Cross War Memorial Children's Hospital ( Site 2601), Cape Town, Western Cape
- Spain (4):
  - Hospital Universitario Sant Joan de Deu ( Site 1704), Esplugues de Llobregat, Barcelona
  - Hospital Infantil Universitario Nino Jesus ( Site 1701), Madrid
  - Hospital Universitario La Paz ( Site 1703), Madrid
  - Hospital Universitario Virgen del Rocio ( Site 1705), Seville
- Sweden (2):
  - ITCC Barnokologen Astrid Lindgrens Barnsjukhus NKS ( Site 1800), Stockholm, Stockholm County
  - Barncancercentrum ( Site 1801), Gothenburg, Västra Götaland County
- United Kingdom (2):
  - Southampton General Hospital ( Site 1900), Southampton, Worcestershire
  - Leeds Teaching Hospitals NHS Trust ( Site 1901), Leeds

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sferra TJ, Merta T, Neely M, Murta de Oliveira C, Lassaletta A, Fortuny Guasch C, Dorr MB, Winchell G, Su FH, Perko S, Fernsler D, Waskin H, Holden SR. Double-Blind, Placebo-Controlled Study of Bezlotoxumab in Children Receiving Antibacterial Treatment for Clostridioides difficile Infection (MODIFY III). J Pediatric Infect Dis Soc. 2023 Jun 30;12(6):334-341. doi: 10.1093/jpids/piad031. PMID 37389891
- See also: Merck Clinical Trial Information — https://merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 148 participants were randomized in the study of which 143 participants received study intervention and were used for safety analysis.
Groups:
- Bezlotoxumab: Participants received 10 mg of bezlotoxumab per kg body weight via a single 60-minute (±10 minutes) intravenous (IV) infusion on Day 1. Additionally, participants received background ABD for 10-21 days per institutional guidelines, at the investigator's discretion.
- Placebo: Participants received placebo for bezlotoxumab consisting of either 0.9% sodium chloride or 5% dextrose via a single 60-minute (±10 minutes) IV infusion on Day 1. Additionally, participants received background ABD for 10-21 days per institutional guidelines, at the investigator's discretion.
Period: Overall Study
Arm/Group | Bezlotoxumab | Placebo
Started | 111 | 37
Treated | 107 | 36
Completed | 103 | 35
Not Completed | 8 | 2
Not completed — Death | 3 | 0
Not completed — Protocol Violation | 4 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bezlotoxumab | Placebo | Total
Number analyzed (Participants) | 111 | 37 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (5.4) | 9.3 (5.3) | 9.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 18 | 69
  Male | 60 | 19 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 9 | 38
  Not Hispanic or Latino | 72 | 27 | 99
  Unknown or Not Reported | 10 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 87 | 32 | 119
  More than one race | 9 | 1 | 10
  Unknown or Not Reported | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve of Bezlotoxumab From Time 0 to Infinity (AUC0-inf)
Description: Blood samples were collected at specified intervals for the determination of AUC0-inf. AUC0-inf was defined as the area under the concentration-time curve of bezlotoxumab from time zero to infinity. Per protocol, AUC0-inf of bezlotoxumab was determined for each age cohort.
Time Frame: Day 1 (2 hours postdose), Days 10, 29, 57, and 85
Population: The analysis population included all participants who received bezlotoxumab, had at least 4 postdose AUC0-inf samples and complied with the protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ug/mL
Groups:
- Bezlotoxumab: Cohort 1 (12 to <18 Years Age): Participants aged 12 to <18 years of age received 10 mg of bezlotoxumab per kg body weight via a single 60-minute (±10 minutes) IV infusion on Day 1. Additionally, participants received background ABD for 10-21 days per institutional guidelines, at the investigator's discretion.
- Bezlotoxumab: Cohort 2 (1 to <12years of Age): Participants aged 1 to <12 years of age received 10 mg of bezlotoxumab per kg body weight via a single 60-minute (±10 minutes) IV infusion on Day 1. Additionally, participants received background ABD for 10-21 days per institutional guidelines, at the investigator's discretion.
Arm/Group | Bezlotoxumab: Cohort 1 (12 to <18 Years Age) | Bezlotoxumab: Cohort 2 (1 to <12years of Age)
Number analyzed (Participants) | 36 | 54
hr*ug/mL | 56100 [49400 to 63700] | 43200 [38900 to 47900]
Statistical Analysis 1: Comparison: Bezlotoxumab: Cohort 1 (12 to <18 Years Age); Test type: Other — The AUC0-inf of bezlotoxumab in Cohort 1 was compared to the AUC0-inf of bezlotoxumab in adults using an analysis of variance (ANOVA) model. The comparison adult PK dataset used was based on participants from 2 adult trials (NCT01241552 and NCT01513239) as a historical control; Geometric Mean Ratio (GMR) = 1.06, 90% CI 2-sided [0.95 to 1.18] — GMR was calculated as the Cohort 1 geometric mean (GM) AUC0-inf / Adult GM AUC0-inf
Statistical Analysis 2: Comparison: Bezlotoxumab: Cohort 2 (1 to <12years of Age); Test type: Other — The AUC0-inf of bezlotoxumab in Cohort 2 was compared to the AUC0-inf of bezlotoxumab in adults using an analysis of variance (ANOVA) model. The comparison adult PK dataset used was based on participants from 2 adult trials (NCT01241552 and NCT01513239) as a historical control; GMR = 0.82, 90% CI 2-sided [0.75 to 0.89] — GMR was calculated as the Cohort 2 GM AUC0-inf / Adult GM AUC0-inf

2. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product and does not imply any judgment about causality. Per protocol, percentage of participants with AEs in the bezlotoxumab and placebo groups were presented.
Time Frame: Up to approximately 12 weeks
Population: The analysis population included all participants who received study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Bezlotoxumab | Placebo
Number analyzed (Participants) | 107 | 36
Percentage of participants | 88.8 | 94.4
Statistical Analysis 1: Comparison: Bezlotoxumab vs Placebo; Test type: Other — Miettinen & Nurminen method was used to generate the estimated difference in percentage and associated 95% confidence intervals (CIs) in bezlotoxumab versus placebo arms; Difference in percentage = -5.7, 95% CI 2-sided [-14.5 to 7.7]

3. Primary Outcome: Percentage of Participants Who Discontinued Study Due to an AE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product and does not imply any judgment about causality. Per protocol, percentage of participants who discontinued study due to AEs in the bezlotoxumab and placebo groups were presented.
Time Frame: Up to approximately 12 weeks
Population: The analysis population included all participants who received study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Bezlotoxumab | Placebo
Number analyzed (Participants) | 107 | 36
Percentage of participants | 0 | 0
Statistical Analysis 1: Comparison: Bezlotoxumab vs Placebo; Test type: Other — Miettinen & Nurminen method was used to generate the estimated difference in percentage and associated 95% CIs in bezlotoxumab versus placebo arms; Difference in percentage = 0.0, 95% CI 2-sided [-9.7 to 3.5]

4. Secondary Outcome: Percentage of Participants Who Had a Clostridium Difficile Infection (CDI) Recurrence
Description: CDI recurrence was defined as diarrhea recurrence (new episode of diarrhea after initial clinical response [ICR] as defined by a change in normal bowel habits for ≥2 days with either watery diarrhea or at least 6 unformed bowel movements [UBMs] within 48-hours) associated with a positive stool test for C. difficile toxin, and for which the participant, in the investigator's opinion, requires and receives ABD treatment for CDI. Per protocol, percentage of participants who had a CDI recurrence in the bezlotoxumab and placebo groups were reported.
Time Frame: Up to approximately 12 Weeks
Population: The analysis population included all participants who received any amount of study intervention, had positive local stool for C. difficile toxin, were taking protocol-defined ABD treatment for CDI on the day of infusion, and achieved an ICR of baseline CDI.
Measure: Number; unit: Percentage of participants
Arm/Group | Bezlotoxumab | Placebo
Number analyzed (Participants) | 98 | 34
Percentage of participants | 11.2 | 14.7
Statistical Analysis 1: Comparison: Bezlotoxumab vs Placebo; Test type: Other — Miettinen and Nurminen method stratified by age cohort (12 to <18 years of age, 1 to <12 years of age) with a Cochran-Mantel-Haenszel weight was used to generate the treatment difference, associated 95% CIs and a 2-sided p-value; p = 0.5701, Stratified Miettinen and Nurminen method; Adjusted difference = -3.7, 95% CI 2-sided [-20.0 to 8.0]

5. Secondary Outcome: Percentage of Participants Who Had a Sustained Clinical Response (SCR)
Description: SCR was defined as the ICR of baseline CDI episode (improvement in number and character of bowel movements and doesn't require further CDI therapy within 2 days after completion of up to 21 days of ABD treatment for CDI) and no CDI recurrence (diarrhea recurrence associated with a positive stool test for C. difficile toxin, and for which the participant, in investigator's opinion, requires and receives ABD for CDI). Per protocol, percentage of participants who had a SCR in bezlotoxumab and placebo groups were presented.
Time Frame: Up to approximately 12 Weeks
Population: The analysis population included all participants who received any amount of study intervention, had positive local stool for C. difficile toxin, and were taking protocol-defined ABD treatment for CDI on the day of infusion.
Measure: Number; unit: Percentage of participants
Arm/Group | Bezlotoxumab | Placebo
Number analyzed (Participants) | 104 | 35
Percentage of participants | 83.7 | 82.9
Statistical Analysis 1: Comparison: Bezlotoxumab vs Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.9165, Stratified Miettinen and Nurminen method; Adjusted difference = 0.8, 95% CI 2-sided [-11.8 to 17.6]

6. Secondary Outcome: Percentage of High-Risk Participants Who Experienced a CDI Recurrence
Description: CDI recurrence was defined as diarrhea recurrence (new diarrhea episode after ICR defined by change in normal bowel habits for ≥2 days with watery diarrhea or at least 6 UBMs within 48-hours) with positive stool test for C. difficile toxin for which participant, in investigator's opinion, requires and receives ABD for CDI. High-risk was meeting ≥1 criteria at/before randomization: a) was immunocompromised b) had ≥1 CDI episode prior to baseline episode c) had severe CDI baseline episode d) had C. difficile ribotype027 in stool at baseline CDI episode e) received ≥1 systemic ABD known to increase CDI risk. Per protocol, percentage of high-risk participants who experienced a CDI recurrence in the bezlotoxumab and placebo groups were presented.
Time Frame: Up to approximately 12 Weeks
Population: The analysis population included all participants who received study intervention, had positive local stool for C. difficile toxin, were taking ABD for CDI on infusion day, achieved ICR of baseline CDI, and were at high-risk of CDI recurrence.
Measure: Number; unit: Percentage of participants
Arm/Group | Bezlotoxumab | Placebo
Number analyzed (Participants) | 91 | 33
Percentage of participants | 12.1 | 15.2
Statistical Analysis 1: Comparison: Bezlotoxumab vs Placebo; Test type: Other — Unstratified Miettinen and Nurminen method was used to generate the treatment difference, associated 95% CIs and a 2-sided p-value; p = 0.6542, Unstratified Miettinen & Nurminen method; Adjusted Difference = -3.1, 95% CI 2-sided [-19.9 to 9.0]

7. Secondary Outcome: Percentage of High-Risk Participants Who Experienced a SCR
Description: SCR was ICR of baseline CDI episode (improvement in number and character of bowel movements and doesn't require further CDI therapy within 2 days after completion of up to 21 days of ABD for CDI) and no CDI recurrence (diarrhea recurrence with positive stool test for C. difficile toxin, for which participant, in investigator's opinion, requires and receives ABD for CDI). High-risk was meeting ≥1 criteria: a) was immunocompromised b) had ≥1 episodes of CDI prior to baseline episode c) had severe CDI baseline episode d) had C. difficile ribotype027 in stool at baseline CDI episode e) received ≥1 systemic ABD known to increase CDI risk. Per protocol, percentage of high-risk participants who had SCR in bezlotoxumab and placebo groups were presented.
Time Frame: Up to approximately 12 Weeks
Population: The analysis population included all participants who received study intervention, had positive local stool for C. difficile toxin, were taking protocol-defined ABD for CDI on the day of infusion, and were at high risk of CDI recurrence.
Measure: Number; unit: Percentage of participants
Arm/Group | Bezlotoxumab | Placebo
Number analyzed (Participants) | 97 | 34
Percentage of participants | 82.5 | 82.4
Statistical Analysis 1: Comparison: Bezlotoxumab vs Placebo; Test type: Other — Unstratified Miettinen and Nurminen method was used to generate treatment difference, associated 95% CIs and a 2-sided p-value; p = 0.9873, Unstratified Miettinen & Nurminen method; Adjusted difference = 0.1, 95% CI 2-sided [-13.0 to 17.4]

8. Secondary Outcome: Percentage of Participants Who Experienced One or More Infusion Related Reaction
Description: Infusion related reaction included events meeting any of the 3 criteria: 1) acute onset of an illness involving skin, mucosal tissue, or both and at least 1 of the following: respiratory compromise, reduced blood pressure (BP) or associated symptoms of end-organ dysfunction 2) two or more of the following after onset of study infusion: involving skin-mucosal tissue, respiratory compromise, reduced BP or associated symptoms, or persistent gastrointestinal symptoms 3) reduced BP after onset of infusion or >30% decrease in systolic BP from baseline. Per protocol, percentage of participants experiencing 1 or more infusion-related reactions within 24 hours following the start of study medication infusion were reported.
Time Frame: Up to approximately 24 hours after infusion on Day 1
Population: The analysis population included all participants who received study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Bezlotoxumab | Placebo
Number analyzed (Participants) | 107 | 36
Percentage of participants | 0.93 | 2.78

9. Secondary Outcome: Percentage of Participants Who Had Positive Antibodies to Bezlotoxumab
Description: Blood samples were collected to determine antibodies to bezlotoxumab. Per protocol, percentage of participants with treatment-emergent positive antibodies to bezlotoxumab following single infusion of bezlotoxumab were reported for each age cohort.
Time Frame: Up to approximately 12 Weeks
Population: The analysis population included all participants who received any amount of bezlotoxumab, had a positive local stool for C. difficile toxin, were taking protocol-defined ABD drug treatment for CDI on the day of infusion, and achieved an ICR of baseline CDI.
Measure: Number; unit: Percentage of participants
Groups:
- Bezlotoxumab: Cohort 2 (1 to <12 Years of Age): Participants aged 1 to <12 years of age received 10 mg of bezlotoxumab per kg body weight via a single 60-minute (±10 minutes) IV infusion on Day 1. Additionally, participants received background ABD for 10-21 days per institutional guidelines, at the investigator's discretion.
Arm/Group | Bezlotoxumab: Cohort 1 (12 to <18 Years Age) | Bezlotoxumab: Cohort 2 (1 to <12 Years of Age)
Number analyzed (Participants) | 44 | 62
Percentage of participants | 2.4 | 1.7

ADVERSE EVENTS:
Time Frame: Up to approximately 14 months
Description: All cause mortality was reported on all randomized participants and non-serious and serious AEs were reported on all participants who received study intervention.
Arm/Group | Bezlotoxumab | Placebo
All-Cause Mortality (participants affected / at risk) | 6/111 | 1/37
Serious Adverse Events (participants affected / at risk) | 57/107 | 29/36
Other Adverse Events (participants affected / at risk) | 65/107 | 28/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bezlotoxumab (N=107) | Placebo (N=36)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 22 (30) | 11 (17)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (6) | 3 (3)
Biliary-bronchial fistula (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Acinetobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Candida sepsis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (2)
Coronavirus infection (Infections and infestations) | 1 (1) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Fungal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis sapovirus (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 3 (3) | 0 (0)
Serratia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 4 (4) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (5) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Vulval cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Venoocclusive disease (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bezlotoxumab (N=107) | Placebo (N=36)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 6 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (8) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 13 (28) | 6 (10)
Constipation (Gastrointestinal disorders) | 7 (11) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 5 (14)
Nausea (Gastrointestinal disorders) | 7 (10) | 4 (5)
Stomatitis (Gastrointestinal disorders) | 8 (10) | 2 (2)
Vomiting (Gastrointestinal disorders) | 14 (16) | 8 (12)
Pyrexia (General disorders) | 15 (22) | 8 (12)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 5 (5) | 2 (4)
Rhinitis (Infections and infestations) | 2 (2) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 9 (12) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 8 (8) | 0 (0)
C-reactive protein increased (Investigations) | 4 (4) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (9) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 15 (22) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Vancomycin infusion reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts and manuscripts regarding this study prior to submission for publication. This will allow the SPONSOR to protect the proprietary information prior to submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT03182907/Prot_SAP_000.pdf